CLINICAL TRIAL: NCT00589186
Title: Phase II Clinical Trial of Tumour Vaccination By Intradermal Delivery of Autologous Dendritic Cells Transduced With Adenoviral Vector (AD5F35) Expressing Latent Membrane Protein-1 (LMP-1) and Latent Membrane Protein-2 (LMP-2) Genes in Combination With Celecoxib in Patient With Metastatic Nasopharyngeal Carcinoma
Brief Title: Vaccine Therapy and Celecoxib in Treating Patients With Metastatic Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000579355; SINGAPORE-NCC-07-11-NPC
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Celecoxib; Flow Cytometry; Immunoenzyme Techniques

INTERVENTIONS:
Biological: Ad5F35-LMP1/LMP2-transduced autologous dendritic cells
Drug: celecoxib
Other: flow cytometry
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus and a person's dendritic cells may help the body build an effective immune response to kill tumor cells. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vaccine therapy together with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with celecoxib works in treating patients with metastatic nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the clinical benefit rate (complete response, partial response, and stable disease for ≥ 14 weeks) in patients with metastatic nasopharyngeal carcinoma treated with autologous dendritic cells (DC) transduced with AD5F35 expressing LMP-1 and LMP-2 when administered in combination with celecoxib.

Secondary

* To evaluate the toxicities of this regimen in these patients.
* To evaluate the specific T-cell response against LMP-1 and LMP-2 as measured by HLA tetramer technology, ELISPOT assay, and delayed-type hypersensitivity in patients treated with this regimen.
* To evaluate the surrogate tumor marker response plasma EBV DNA by real-time PCR in these patients.
* To evaluate and characterize immunological cell types and tumor characteristics in biopsy specimens of patients treated with this DC vaccine and compare it with pre-vaccine biopsy specimens.
* To evaluate progression-free survival and overall survival of patients who show initial clinical benefit to DC vaccine.

OUTLINE: Patients undergo blood collection for the preparation of the autologous dendritic cell (DC) vaccine. Immature DCs are transduced with latent membrane protein-1 (LMP-1) and latent membrane protein-2 (LMP-2) using the adenoviral vector 5F35. Beginning 1 week after blood collection, patients receive vaccination with autologous DCs transduced with AD5F35-LMP-1/LMP-2 intradermally every 2 weeks for a total of 5 vaccinations. Patients also receive celecoxib twice a day beginning 1 week before the first vaccination and continuing for up to 6 weeks after completion of the last vaccination.

Patients who demonstrate clinical benefit after completion of 5 courses of vaccination may continue to receive the DC vaccine alone off study every 2 weeks until disease progression (based on CT scan findings) or at the investigator's discretion.

Patients undergo blood and tumor tissue sample collection periodically for laboratory studies. Blood samples are analyzed using MHC tetramer analysis; enzyme-linked immunospot (ELISPOT) analysis; EBV DNA titers to assess response; and flow cytometry to assess lymphocyte kinetics. Tumor tissue samples are used for immunological studies. Delayed-type hypersensitivity is also assessed.

After completion of study treatment, patients are followed monthly for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nasopharyngeal carcinoma (NPC)

  * Metastatic disease
  * WHO type II/III disease
* Measurable disease
* Meets 1 of the following criteria:

  * Progression on one or more lines of polychemotherapy for treatment of metastatic disease
  * Failed non-myeloablative hematopoietic stem cell transplant
* No active CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Hemoglobin ≥ 8.5 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal
* ALT or AST ≤ 5 times normal
* Creatinine clearance ≥ 40 mL/min
* Left ventricular ejection fraction ≥ 45% by MUGA
* Corrected DLCO > 50% of predicted
* No active or prior gastrointestinal bleeding
* No history of adverse reaction to NSAIDs or sensitivity to celecoxib
* No cardiac disease, including any of the following:

  * Symptomatic congestive heart failure
  * Active angina pectoris
  * High-risk uncontrolled arrhythmia
  * Uncontrolled hypertension
* No pulmonary disease, including any of the following:

  * Severe chronic obstructive lung disease
  * Uncontrolled large pleural effusion
  * Severe restrictive lung disease
* No cerebrovascular accident
* No transient ischemic attack
* No HIV positivity
* No active uncontrolled infection
* No symptomatic leukoencephalopathy or other neuropsychiatric abnormalities
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior celecoxib allowed
* At least 28 days since prior chemotherapy
* At least 100 days since prior non-myeloablative hematopoietic stem cell transplant
* At least 2 months since prior donor lymphocyte infusions
* More than 28 days since prior participation in another clinical trial with any investigational drugs
* No other concurrent experimental drugs
* No other concurrent anticancer therapy
* No concurrent anticoagulation with warfarin or low molecular weight heparin
* No other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) or aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) (complete response [CR], partial response [PR], and stable disease [SD] for ≥ 14 weeks) as defined by RECIST criteria

SECONDARY OUTCOMES:
Response rate (CR and PR)
Overall survival
Progression-free survival
Toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Toh Han Chong, MD, MBBS, MRCP, Study Chair — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore